CLINICAL TRIAL: NCT06617676
Title: Transcutaneous Tibial Nerve Stimulation for Overactive Bladder Syndrome and Associated Gait Changes in Post-menopausal Women
Acronym: TTNS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, Amanda Mahoney, Clinical Assistant Professor - Physical Therapy, Louisiana State University Health Sciences Center Shreveport
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002713
Record Dates: First submitted 2024-09-26; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Overactive Bladder Syndrome; Urinary Incontinence, Urge; Nocturia
Keywords: Overactive bladder syndrome; Transcutaneous sacral nerve stimulation; Falls; Urinary urgency; Urinary frequency; Nocturia
MeSH Terms: conditions — Urinary Incontinence, Urge; Nocturia

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of of the three groups in parallel for the duration of the study. The variable in the intervention will be the number of treatments they receive per week.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TTNS - two times per week (Experimental): Participants will receive transcutaneous tibial nerve stimulation for 30 minutes with a frequency of 12 Hz, pulse width of 300 microseconds, and to an intensity of the participant's tolerance under the motor threshold. This group will receive treatment two times per week.
  Interventions: Device: Transcutaneous tibial nerve stimulation
- TTNS - four times per week (Experimental): Participants will receive transcutaneous tibial nerve stimulation for 30 minutes with a frequency of 12 Hz, pulse width of 300 microseconds, and to an intensity of the participant's tolerance under the motor threshold. This group will receive treatment four times per week.
  Interventions: Device: Transcutaneous tibial nerve stimulation
- No treatment group (No Intervention): Treatment will be deferred after 12 weeks.

INTERVENTIONS:
Device: Transcutaneous tibial nerve stimulation — Two electrodes will be place over the tibial nerve over the medial ankle. The electrical stimulation will be turned up to patient tolerance at a sensory level only.
  Arms: TTNS - four times per week; TTNS - two times per week

SUMMARY:
The goal of this clinical trial is to learn if surface tibial electrical stimulation (mild electrical signals on the inside of the ankle) helps women 60 years or older with urine leakage that happens on the way to the bathroom or at night time. The main questions it aims to answer are: 1). How many treatments per week over a 12-week period improve a person's bladder symptoms?; 2). Is a person more confident that they will not fall and / or leak urine on the way to the bathroom after the treatment with the electrical stimulation treatments; 3). Does the way a person walks when they need to go to the bathroom change after they have had the electrical stimulation? They will visit the clinic 3 times to complete several questionnaires and walk with a full bladder and empty bladder. On the first visit, the participant will be taught how to use the electrical stimulation device. Participants will either receive the treatment 2 or 4 times per week for 12 weeks or no treatment with the option to receive treatment following the 12 weeks. Participants will be given a bladder diary to complete at the start of treatment, at 6 weeks, then at 12 weeks and will be instructed in completion. They will drink water until they have a strong urge to urinate, then will walk along an electronic pathway and will go empty their bladder. After emptying, they will walk back along the electronic pathway again. They will also complete a Timed Up and Go test - stand up from a chair, walk 3 meters, then turn around, walk back, then sit down. At the 6th week follow up and the 12th week follow up, they will complete each questionnaire again and complete the walking tasks again.

DETAILED DESCRIPTION:
This study will improve standardization for the delivery of transcutaneous tibial nerve stimulation as a treatment modality for overactive bladder in post-menopausal women and contribute to lower cost care options within the home environment. This is a prospective randomized control trial where the participants' baseline conditions will be utilized for comparison with post-treatment. The independent variable is transcutaneous tibial nerve stimulation. The dependent variables are urinary frequency and urinary continence episodes based on three-day bladder diary, OAB-V8, Overactive Bladder Symptom Severity Score (OABSS), Activities-specific Balance Confidence Scale (ABC-16), Geriatric Self-efficacy Index for Urinary Incontinence (GSE-UI), and the Timed-Up and Go test (TUGT). Additional pre- and post- test variables that will be considered are spatiotemporal measurements of gait with both full and empty bladder conditions.

At the first session at the School of Allied Health Professions following screening and consent, participants will complete the OAB-SS, ABC-16, and the GSE-UI. Participants will be asked to start drinking water at the start of the first session. Once the participant notes a strong desire to void that is difficult to defer based on the urgency severity scale (USS), the participant will walk along the GaitRITE pathway to the restroom. Participant will void into a urine specimen collector and bladder volume will be recorded, but urine will not be retained. The participant will then walk back over the electronic pathway to collect empty bladder condition gait. Participant will then complete the TUGT. Following this testing, participants will be instructed in home use of the transcutaneous tibial nerve stimulation. Participants will place one electrode 3 finger widths above the medial malleolus with the other placed below the medial malleolus with the following parameters: 10 Hertz, 200 microseconds, for 30 minutes to a strong but comfortable level that is under the motor threshold. Participants will complete these sessions either two or four times per week for 12 weeks or will receive no treatment for the 12 weeks. Participants will be given a log for home use to document their compliance with the home treatment.

Participants will follow up at the School of Allied Health Professions at the 6-week mark to complete the gait testing and Activities-specific Balance Confidence Scale and the Geriatric Self-Efficacy Index for Urinary Incontinence. Participants will be given supplies to complete an additional three-day bladder diary to bring with them for the 12-week follow-up. Following 12 weeks of transcutaneous tibial nerve stimulation, participants will return to the School of Allied Health Professions to complete the procedure described above.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria include females over 60 years of age who score an 8 or greater on the OAB-V8 with no exclusion criteria.

-

Exclusion Criteria: those who experience stress UI only, have a pacemaker, neurologic deficit (e.g. Parkinson's disease, multiple sclerosis, spinal cord injury), current urinary tract infection, known active cancer, or current OAB medication use (Tolterdine, etc.) with consideration of a washout period, and inability to walk 30 meters.

-

Ages: 60 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender females, biological females
Enrollment: 60 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Overactive Bladder Symptom Score (OABSS) | From enrollment to the end of treatment at 12 weeks
  Overactive Bladder Symptom Score is a self-reported outcome measure that will be collected at multiple time frames - initial day, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, and 12 weeks.

SECONDARY OUTCOMES:
Geriatric Self-efficacy Index for Urinary Incontinence | From enrollment to the end of treatment at 12 weeks
  The Geriatric Self-efficacy Index for Urinary Incontinence is a self-reported outcome measure that will be completed at the initial clinic visit, 6-week follow up clinic visit, 12-week follow up clinic visit.
Activities-specific Balance Confidence Scale | From enrollment to the end of treatment at 12 weeks
  The Activities-specific Balance Confidence Scale is a self-reported outcome measure that will be completed at the initial clinic visit, 6-week follow up clinic visit, 12-week follow up clinic visit.
Timed Up and Go Test | From enrollment to the end of treatment at 12 weeks
  The Timed Up and Go Test is a walking test that will be performed at the initial clinic visit, 6-week follow up clinic visit, 12-week follow up clinic visit. Participants will rise from a chair, walk three meters, turn around, walk back to the chair, and sit back down for time.
Ambulation with a strong desire to void | From enrollment to the end of treatment at 12 weeks
  Participants will drink water until they reach the sensation of a strong desire to void. They will walk across an electronic pathway to determine gait velocity, step length, and step width. They will complete this at the initial clinic visit, 6-week follow up clinic visit, and 12-week follow up clinic visit.
Ambulation with empty bladder conditions | From enrollment to the end of treatment at 12 weeks
  Participants will walk across an electronic pathway after emptying their bladder to determine gait velocity, step length, and step width. They will complete this at the initial clinic visit, 6-week follow up clinic visit, and 12-week follow up clinic visit.
Three Day Bladder Diary | From enrollment to the end of treatment at 12 weeks
  Participants will complete a three day voiding diary to determine urinary frequency, urinary urgency, and the number of nighttime voids. These will be completed at the initial clinic visit, 6-week follow up clinic visit, and 12-week follow up clinic visit.

IPD SHARING:
Plan to Share IPD: No